CLINICAL TRIAL: NCT04963517
Title: 3D Gait Analysis to Determine Functional Limitations and Evaluate a Training Intervention in Young People with Tumor Endoprosthesis of the Lower Extremity
Brief Title: Exercise Intervention for Bone Tumor Patients
Acronym: proGAIT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Miriam Götte, Principal investigator, Head of exercise oncology group, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: proGAIT
Record Dates: First submitted 2021-06-15; First posted 2021-07-15 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Bone Sarcoma
Keywords: exercise; lower limb endoprosthesis; pediatric oncology; gait quality; 3D gait analysis
MeSH Terms: conditions — Bone Neoplasms; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise therapy (Experimental): 8 weeks personalized, multi-modal exercise with focus on lower extremity
  * Initial consultation with recommendations for general physical activity
  * Brochure with exercise recommendations
  * 2x per week multi-modal group-based and supervised exercise (endurance, strength, mobility, coordination)
  * week 1 and 2 supervised, week 3 and 4 partially supervised, week 5 and 6 only one supervised session, week 7 and 8 last two sessions supervised
  Interventions: Behavioral: Exercise therapy
- Information group (Active Comparator): * Initial consultation with recommendations for general physical activity
  * Brochure with exercise recommendations.
  Interventions: Other: Information

INTERVENTIONS:
Behavioral: Exercise therapy — 8 weeks personalized, multi-modal exercise with focus on lower extremity
  Other Names: physical activity intervention
  Arms: Exercise therapy
Other: Information — * Initial consultation with recommendations for general physical activity
  * Brochure with exercise recommendations.
  Arms: Information group

SUMMARY:
The proGait-study is a two-arm exercise intervention study for AYA-patients with lower extremity tumor endoprosthesis in the follow-up care. This clinical trial will investigate the effects of an 8-week personalized multi-modal exercise intervention of lower extremity muscles on gait quality in adolescents and young adults with cancer diagnosis beginning at least 12 months after endoprosthesis implantation.

DETAILED DESCRIPTION:
The main objective of the proGait-study is to investigate the effects of an 8-week personalized, partially supervised exercise program for lower extremity muscles on gait kinematics of adolescents and young adults, who are in follow-up care after cancer treatment and at least 12 months after endoprosthesis implantation. This randomized controlled trial will include n=20-30 patients. Patients will be randomly assigned to the intervention or control group. Patients in the intervention group will perform two supervised exercise sessions in week one and two. In the following weeks, they will perform in a mix of supervised and unsupervised exercise sessions to introduce the patients into independent exercise. Both groups receive recommendations for individual lower extremity exercise. Secondary aims of this interventional study are to evaluate functional mobility, knee range of motion and patient-reported outcomes including QoL and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults between 15 and 45 years of age
* Completion of acute cancer treatment and receiving follow-up care in Essen (University Hospital Essen)
* At least 12 months post endoprosthesis implantation
* Signed informed consent (Parents and Patient)

Exclusion Criteria:

* <15 years of age, >45 years of age
* time post implantation <12 months
* Medical condition that limits participation in one of the study arms
* Inability to follow the training-protocol

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2021-08-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Gait Profile Score | 8 weeks
  Marker based 3D gait analysis is performed on a 15m runway and recorded at 120Hz with 8 cameras from different projection angles around the runway (Vicon, Oxford, UK). Gait Profile Score is based on the averaged RMS differences in lower body kinematics (Pelvis tilt ant/post, Pelvis tilt up/down, Pelvis internal rotation/external rotation, Hip joint flexion/extension, Hip joint adduction/abduction, Hip joint internal rotation/external rotation, Knee flexion/extension, Ankle joint Dorsiflexion/Plantarflexion, Foot opening angle Internal rotation/External rotation) of subjects and kinematic reference data from a healthy population during a time normalized gait cycle. A lower GPS would indicate less deviation from a healthy populations gait pattern and thus indicate a better outcome.

SECONDARY OUTCOMES:
Functional Mobility | 8 weeks
  Functional Mobility Assessment score (points, score range 0 - 70, higher score = better outcome) between both study arms from T0 to T1
Subjective functional outcome | 8 weeks
  Change in Musculoskeletal Tumor Society Score (questionnaire score, score range 0 - 30, higher score = better outcome) between both study arms
Subjective functional measure | 8 weeks
  Change in Toronto Extremity Salvage Score(questionnaire score, score range 0 - 100, higher score = better outcome) between both study arms
Subjective Quality of Life Adults | 8 weeks
  Change in Quality of Life (QLQ-C30 questionnaire score from 0 - 100) between both study arms
Subjective Quality of Life Adolescents | 8 weeks
  Change in Quality of Life (PedsQL cancer module, questionnaire score from 0 - 100) between both study arms
Fatigue Adults | 8 weeks
  Change in Fatigue (EORTC QLQ Fatigue questionnaire range 0 - 100, higher score = worse outcome) between both study arms
Range of motion | 8 weeks
  Change in affected knee range of motion (angular degree °) assessed with goniometry between both study arms
Gait kinematics | 8 weeks
  Changes in lower body gait kinematics between both study arms from T0 to T1 by assessing the Gait Deviation Index (GDI), measure of difference between subjects and a healthy control dataset of lower body kinematics. A GDI of 100 indicates a subject whose gait is at least as close to the healthy average as that of a randomly selected healthy individual. Thus, a GDI of 100 or higher indicates the absence of gait pathology. Every 10 points that the GDI falls below 100 corresponds one standard deviation away from the healthy populations mean.
Fatigue Adolescents | 8 weeks
  Change in Fatigue (PedsQL fatigue questionnaire score, range 0 - 100, higher score = worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Götte, PhD, Principal Investigator — University Hospital, Essen
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basteck S, Guder WK, Dirksen U, Krombholz A, Streitburger A, Reinhardt D, Gotte M. Effects of an Exercise Intervention on Gait Function in Young Survivors of Osteosarcoma with Megaendoprosthesis of the Lower Extremity-Results from the Pilot Randomized Controlled Trial proGAIT. Curr Oncol. 2022 Oct 14;29(10):7754-7767. doi: 10.3390/curroncol29100613. PMID 36290890